CLINICAL TRIAL: NCT06486233
Title: Comparison of Mortality and Complication Rates (Re-myocardial Infarction, Heart Failure, Re-hospitalization, Stroke) After 12 Months Between Two Groups of Patients Undergoing Early Invasive and Late Invasive Strategies in Patients With Elderly Patients With High - Risk Non-ST-segment Elevation Acute Coronary Syndrome.
Brief Title: Studying the Effectiveness of Early Invasive Treatment in Elderly Patients With High-risk Non-ST-segment Elevation Acute Coronary Syndrome.
Status: Recruiting | Type: Observational
Sponsor: Gia Dinh People Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 329/HDDD-DHYD
Record Dates: First submitted 2024-06-12; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Myocardial Infarction
Keywords: percutaneous coronary intervention, elderly, non-ST-segment Elevation
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Observe the patient with early percutaneous coronary intervention: Elderly patients with non-ST-segment elevation acute coronary syndrome receive early percutaneous coronary intervention (< 24 hours after diagnosis).
- Observe the patient with late percutaneous coronary intervention: Elderly patients with non-ST elevation acute coronary syndrome undergoing late percutaneous coronary intervention (≥ 24 hours after diagnosis)

SUMMARY:
The goal of this is observational study is to compare about MACE events and predisposing factors related to MACE events in elderly patients with high-risk non-ST acute coronary syndromes receiving early versus late invasive treatment . This study will anwser two questions.

Question 1: What will factors associate with implementing a late invasive strategy in elderly patients with high-risk non-ST-segment elevation acute coronary syndrome ? Question 2: Is a meaningful difference about mortality and complication rates as re-myocardial infarction, heart failure, re-hospitalization, stroke after 12 months between two groups of patients undergoing early invasive and late invasive strategies in elderly patients with in high-risk non-ST-segment elevation acute coronary syndrome?

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years and older
* high - risk non-ST-segment elevation acute coronary syndrome (according to the 2023 European Heart Association recommended standards).
* receives reperfusion intervention.

Exclusion Criteria:

* Acute coronary syndrome due to stent thrombosis, or coronary artery bypass graft occlusion.
* Incomplete medical records.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 60 years and older were diagnosed with non-ST elevation acute coronary syndrome. Diagnosed with high-risk acute non-ST elevation syndrome and treated at Gia Dinh People's Hospital, Thong Nhat Hospital during the study period.
Sampling Method: Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital death | one month
  recorded when death occurs during treatment or is confirmed by in-hospital monitoring

SECONDARY OUTCOMES:
after 12 months death | one year
  determined by the patient follow-up period from hospital discharge until results were recorded
MACE after 12 months include re-admission, recurrent myocardial infarction , stroke, heart failure | one year
  recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Gia Dinh people hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No